CLINICAL TRIAL: NCT01992926
Title: Facilitating Anemia Treatment Risk Communication for Patients With Kidney Disease: Decision Aid Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Kerri Cavanaugh, Assistant Professor, Vanderbilt University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 130784
Record Dates: First submitted 2013-11-14; First posted 2013-11-25 (Estimated); Last update posted 2015-01-22 (Estimated); Status verified 2015-01

CONDITIONS: Chronic Kidney Disease; End Stage Renal Disease
Keywords: health literacy; health numeracy
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- interactive educational intervention (Active Comparator): Physicians will use an interactive educational worksheet during the standard-of-care clinic visit.
  Interventions: Behavioral: interactive educational intervention
- control group (No Intervention): Physicians will conduct the standard-of-care clinic visit as usual.

INTERVENTIONS:
Behavioral: interactive educational intervention — Use of a concise, literacy-sensitive, physician-led, educational interaction with the patient.
  Arms: interactive educational intervention

SUMMARY:
Anemia is a common complication of chronic kidney disease (CKD). In anemia of chronic kidney disease, patients suffer from low hemoglobin levels, which contribute to feelings of malaise and fatigue. The current accepted practice is often to administer erythropoietin-stimulating agents (ESAs), which act like the body's natural hormones to stimulate the production of red blood cells from bone marrow. Although ESAs are widely used in CKD, recent evidence suggests that they are not as safe as previously thought. In this study, we seek to test a decision aid to be used when a patient visits his or her nephrologist at Vanderbilt. The objective of the decision aid is to reduce patient confusion, improve their satisfaction with their care, improve their knowledge of kidney disease, and ultimately bring more clarity to patients about a controversial but ubiquitous drug.

The decision aid will be about 1 page long and will include questions and information that might help the patient be more active and informed regarding the choice of a course of ESA therapy. We will ask patients to answer questions before and after their clinic visits regarding their satisfaction and confidence in their treatment and their knowledge of kidney disease; we will ask some of the same questions 3 months after the clinic visit. We will compare patients who are counseled using the decision aid to patients who are not. We anticipate total experiment running time to be approximately 5 months to recruit and follow up on all patients.

ELIGIBILITY:
Inclusion Criteria:

* Has Chronic Kidney Disease or End Stage Renal Disease
* Over 18, under 80 years of age
* Currently receiving care in the Vanderbilt Nephrology or Dialysis Clinics
* Receiving ESAs for anemia
* Speaks and can read English (no previous use of interpreter services)
* No significant visual impairment documented in medical record

Exclusion Criteria:

* Diagnosed cognitive disability
* Stated inability to converse and read fluently in English, or prior use of translation services
* Poor visual acuity

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2013-11; Primary Completion 2014-08 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
change in patient understanding of anemia and treatment options | baseline and 3 months
  Change from baseline in the following surveys/questionaires at 3 months:
  * Anemia Knowledge Survey (PAKKD)
  * Perceived Kidney Self-Management Scale (PKiSMS or PDiSMS for ESRD)
  * Social Support Measure (MSPSS)
  * Perceived Efficacy in Patient-Physician Interactions (PEPPI)

CONTACTS AND LOCATIONS:
Overall Officials: Kerri Cavanaugh, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Beach LB, Wild M, Ramachandran G, Ikizler HO, Cavanaugh KL. Protocol of a randomized controlled trial of an erythropoietin stimulating agent decision aid for anemia treatment in kidney disease. BMC Nephrol. 2016 Jul 18;17(1):86. doi: 10.1186/s12882-016-0301-z. PMID 27430294